CLINICAL TRIAL: NCT05280782
Title: Development and Translation of Generator-Produced PET Tracer for Myocardial Perfusion Imaging
Brief Title: Development and Translation of Generator-Produced PET Tracer for Myocardial Perfusion Imaging-Dosimetry Group
Acronym: GALMYDAR
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pamela Woodard, MD, H M Wilson Professor of Radiology, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202107042; IND 157468 (Other: U.S. Food and Drug Administration); R01HL142297 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-03-15 (Actual); Results first posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Coronary Artery Disease
Keywords: myocardial perfusion imaging; pharmacological stress; biodistribution; positron emission tomography; myocardial blood flow
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosimetry Group (Experimental): Normal Volunteers will receive a single intravenous injection of 8 mCi ± 20% (6.4-9.6 mCi) of the PET radiotracer 68Ga-Galmydar. They will undergo whole-body PET/CT imaging at three-time points, immediately post [68Ga]Galmydar injection, and at 2 hours and 4 hours after injection. Serum chemistries, complete blood count, EKG, vital signs, and physical examination will performed before injection and at the completion of the examinations.
  Interventions: Drug: Ga-68 Galmydar

INTERVENTIONS:
Drug: Ga-68 Galmydar — Single intravenous injection of the PET radiotracer 68Ga-Galmydar.
  Other Names: IND 157468

SUMMARY:
This study is a single center, early phase 1 clinical imaging study designed to assess the dosimetry of 68Ga-Galmydar for PET/CT imaging.

DETAILED DESCRIPTION:
The objective is to evaluate dosimetry, biodistribution, safety, and imaging characteristics following a single 68Ga-Galmydar injection in normal healthy volunteers. Healthy adult normal volunteers (n=8, 4 males; 4 females) will undergo whole-body imaging (dosimetry group).

Healthy adult normal volunteers (n=8, 4 males; 4 females) will receive a single intravenous Ga-68 Galmydar administration of 8 mCi ± 20% (6.4-9.6 mCi) with a mass of ≤ 10 µg followed by whole-body PET/CT imaging.

ELIGIBILITY:
Inclusion Criteria:

• Healthy men and women, 18-99 years of age and any race

Exclusion Criteria:

* Inability to receive and sign informed consent;
* Positive urine screen for drugs of abuse at screening or before dosing or over-the- counter drug use or herbal preparations within the 2-week period prior to enrollment;
* Participation in another research study with a study drug, including a diagnostic or therapeutic radiopharmaceutical, to be administered during this study or which was or will be administered within 10 hall-lives of the radiopharmaceutical.
* Severe claustrophobia;
* Pregnant or breastfeeding.
* Body mass index < 18 kg/m2 or > 40 kg/m2.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Woodard, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sivapackiam J, Laforest R, Sharma V. 68Ga[Ga]-Galmydar: Biodistribution and radiation dosimetry studies in rodents. Nucl Med Biol. 2018 Apr;59:29-35. doi: 10.1016/j.nucmedbio.2017.11.008. Epub 2017 Dec 1. PMID 29454148

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dosimetry Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 79.4 (18.3)

OUTCOME MEASURES:

1. Primary Outcome: Organ Dosimetry
Description: On whole body PET/CT, regions of interest are drawn on the liver, spleen, kidney, lumbar vertebrae and left ventricle of the heart. Average organ dose is measured and compared. Organ radiation dose is measured and reported in rad/mCi.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Mean (Standard Deviation); unit: rad/mCi
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
rad/mCi
  Adrenals | 0.109 (0.015)
  Brain | 0.019 (0.007)
  Breasts | 0.012 (0.014)
  Esophagus | 0.034 (0.008)
  Eyes | 0.018 (0.007)
  Gallbladder Wall | 1.923 (1.134)
  Left Colon | 0.107 (0.037)
  Small Intestine | 0.405 (0.181)
  Stomach Wall | 0.037 (0.008)
  Right Colon | 0.327 (0.157)
  Rectum | 0.037 (0.007)
  Heart Wall | 0.110 (0.026)
  Kidneys | 0.483 (0.197)
  Liver | 0.364 (0.039)
  Lungs | 0.032 (0.008)
  Ovaries | 0.042 (0.009)
  Pancreas | 0.046 (0.024)
  Salivary Glands | 0.378 (0.554)
  Red Marrow | 0.064 (0.021)
  Osteogenic Cells | 0.041 (0.010)
  Spleen | 0.246 (0.055)
  Thymus | 0.022 (0.010)
  Thyroid | 0.098 (0.091)
  Urinary Bladder Wall | 0.137 (0.018)
  Uterus | 0.066 (0.031)
  Total Body | 0.045 (0.007)

2. Primary Outcome: Biodistribution
Description: The organ with the highest radiation dose in rad/mCi is determined to be the dose-critical organ. The organ showing the largest dose is the gallbladder wall.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Mean (Standard Deviation); unit: rad/mCi
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
rad/mCi | 1.923 (1.134)

3. Primary Outcome: Total Effective Dose of the Radiotracer
Description: Total Effective Dose of the radiotracer is calculated using ICRP-60 organ weights and is reported in rem/mCi.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Mean (Standard Deviation); unit: rem/mCi
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
rem/mCi | 0.103 (0.012)

4. Secondary Outcome: Clinically Significant Change in Blood Pressure.
Description: The following variables are considered clinically significant if changes occur from baseline. A systolic BP of < 90 or > 160 mmHg or a diastolic BP of < 50 or > 100 mmHg or a 20 mmHg change from baseline in the SBP or DBP.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Systolic Blood Pressure: Normal | 8
  Baseline Systolic Blood Pressure: Abnormal | 0
  Post-Injection Systolic Blood Pressure: Normal | 8
  Post-Injection Systolic Blood Pressure: Abnormal | 0
  Baseline Diastolic Blood Pressure: Normal | 8
  Baseline Diastolic Blood Pressure: Abnormal | 0
  Post-Injection Diastolic Blood Pressure: Normal | 8
  Post-Injection Diastolic Blood Pressure: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Systolic Blood Pressure values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Systolic Blood Pressure values were normal
Statistical Analysis 2: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Diastolic Blood Pressure values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Diastolic Blood Pressure values were normal

5. Secondary Outcome: Clinically Significant Change in Heart Rate.
Description: A heart rate of < 50 BPM or > 100 or a 20 BPM change from baseline.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Heart Rate: Normal | 8
  Baseline Heart Rate: Abnormal | 0
  Post-Injection Heart Rate: Normal | 8
  Post-Injection Heart Rate: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Heart Rate values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Heart Rate values were normal

6. Secondary Outcome: Clinically Significant Change in Respiratory Rate.
Description: A respiratory rate of < 12 or > 20 breaths/min.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Respiratory Rate: Normal | 8
  Baseline Respiratory Rate: Abnormal | 0
  Post-Injection Respiratory Rate: Normal | 7
  Post-Injection Respiratory Rate: Abnormal | 1
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Respiratory Rate values. The values were categorized as Normal or Abnormal; p = 0.016, McNemar — The threshold for statistical significance was p = 0.05

7. Secondary Outcome: Clinically Significant Elevation in Oral Temperature
Description: Oral temperature of >100 degrees F.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Temperature: Normal | 8
  Baseline Temperature: Abnormal | 0
  Post-Injection Temperature: Normal | 8
  Post-Injection Temperature: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Temperature values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Temperature values were normal

8. Secondary Outcome: Clinically Significant Change in EKG Showing New AV Block
Description: A change in EKG showing new AV Block (Type 1 or Type 2), Mobitz 2:1, or QTc ≥ 500ms).
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline EKG: Normal | 8
  Baseline EKG: Abnormal | 0
  Post-Injection EKG: Normal | 8
  Post-Injection EKG: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection EKG. The outcomes were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the EKGs were normal

9. Secondary Outcome: Clinically Significant Change in EKG Showing New Bradycardia
Description: New heart rate < 40 BPM.
Time Frame: 6 hours from 68Ga-Galmydar injection
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline EKG: Normal | 8
  Baseline EKG: Abnormal | 0
  Post-Injection EKG: Normal | 8
  Post-Injection EKG: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — [test comment as in outcome 8, analysis 1]; [other analysis details as in outcome 8, analysis 1]

10. Secondary Outcome: Clinically Significant Change in Serum Chemistries: Sodium, Potassium, Chloride, CO2
Description: Serum chemistries (sodium, potassium, chloride, CO2) measured in mmol/L. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: All patients were scheduled to undergo serum chemistries. Three patients did not undergo post-injection serum chemistries due to various issues (IV, blood hemolysis, or wrong labs).
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Sodium: Normal | 8
  Baseline Sodium: Abnormal | 0
  Post-Injection Sodium: number analyzed (Participants) | 5
  Post-Injection Sodium: Normal | 5
  Post-Injection Sodium: Abnormal | 0
  Baseline Potassium: Normal | 8
  Baseline Potassium: Abnormal | 0
  Post-Injection Potassium: number analyzed (Participants) | 5
  Post-Injection Potassium: Normal | 5
  Post-Injection Potassium: Abnormal | 0
  Baseline Chloride: Normal | 8
  Baseline Chloride: Abnormal | 0
  Post-Injection Chloride: number analyzed (Participants) | 5
  Post-Injection Chloride: Normal | 5
  Post-Injection Chloride: Abnormal | 0
  Baseline CO2: Normal | 7
  Baseline CO2: Abnormal | 1
  Post-Injection CO2: number analyzed (Participants) | 5
  Post-Injection CO2: Normal | 5
  Post-Injection CO2: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Sodium values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Sodium values were normal
Statistical Analysis 2: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Potassium values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Potassium values were normal
Statistical Analysis 3: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Chloride values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Chloride values were normal
Statistical Analysis 4: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection CO2 values. The values were categorized as Normal or Abnormal; p = 0.219, McNemar — The threshold for statistical significance was p = 0.05

11. Secondary Outcome: Clinically Significant Change in Serum Chemistries: Glucose, Calcium Creatinine, BUN, Total Bilirubin
Description: Serum chemistries (glucose, calcium creatinine, BUN, total bilirubin), measured in mg/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Glucose: Normal | 7
  Baseline Glucose: Abnormal | 1
  Post-Injection Glucose: number analyzed (Participants) | 5
  Post-Injection Glucose: Normal | 4
  Post-Injection Glucose: Abnormal | 1
  Baseline Calcium: Normal | 7
  Baseline Calcium: Abnormal | 1
  Post-Injection Calcium: number analyzed (Participants) | 5
  Post-Injection Calcium: Normal | 4
  Post-Injection Calcium: Abnormal | 1
  Baseline Creatinine: Normal | 6
  Baseline Creatinine: Abnormal | 2
  Post-Injection Creatinine: number analyzed (Participants) | 5
  Post-Injection Creatinine: Normal | 5
  Post-Injection Creatinine: Abnormal | 0
  Baseline BUN: Normal | 8
  Baseline BUN: Abnormal | 0
  Post-Injection BUN: number analyzed (Participants) | 5
  Post-Injection BUN: Normal | 4
  Post-Injection BUN: Abnormal | 1
  Baseline Total Bilirubin: Normal | 7
  Baseline Total Bilirubin: Abnormal | 1
  Post-Injection Total Bilirubin: number analyzed (Participants) | 5
  Post-Injection Total Bilirubin: Normal | 5
  Post-Injection Total Bilirubin: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Glucose values. The values were categorized as Normal or Abnormal; p = 0.375, McNemar — The threshold for statistical significance was p = 0.05
Statistical Analysis 2: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Calcium values. The values were categorized as Normal or Abnormal; p = 0.375, McNemar — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Creatinine values. The values were categorized as Normal or Abnormal; p = 0.453, McNemar — The threshold for statistical significance was p = 0.05
Statistical Analysis 4: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection BUN values. The values were categorized as Normal or Abnormal; p = 0.125, McNemar — The threshold for statistical significance was p = 0.05
Statistical Analysis 5: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Total Bilirubin values. The values were categorized as Normal or Abnormal; p = 0.219, McNemar — The threshold for statistical significance was p = 0.05

12. Secondary Outcome: Clinically Significant Change in Serum Chemistries: Total Protein, Albumin.
Description: Serum chemistries (total protein, albumin), measured in g/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Total Protein: Normal | 8
  Baseline Total Protein: Abnormal | 0
  Post-Injection Total Protein: number analyzed (Participants) | 5
  Post-Injection Total Protein: Normal | 5
  Post-Injection Total Protein: Abnormal | 0
  Baseline Albumin: Normal | 7
  Baseline Albumin: Abnormal | 1
  Post-Injection Albumin: number analyzed (Participants) | 5
  Post-Injection Albumin: Normal | 5
  Post-Injection Albumin: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Total Protein values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Total Protein values were normal
Statistical Analysis 2: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Albumin values. The values were categorized as Normal or Abnormal; p = 0.219, McNemar — The threshold for statistical significance was p = 0.05

13. Secondary Outcome: Clinically Significant Change in Serum Chemistries: Alkaline Phosphatase, ALT, AST
Description: Serum chemistries (alkaline phosphatase), measured in U/L. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Alkaline Phosphatase: Normal | 8
  Baseline Alkaline Phosphatase: Abnormal | 0
  Post-Injection Alkaline Phosphatase: number analyzed (Participants) | 5
  Post-Injection Alkaline Phosphatase: Normal | 5
  Post-Injection Alkaline Phosphatase: Abnormal | 0
  Baseline ALT: Normal | 7
  Baseline ALT: Abnormal | 1
  Post-Injection ALT: number analyzed (Participants) | 5
  Post-Injection ALT: Normal | 5
  Post-Injection ALT: Abnormal | 0
  Baseline AST: Normal | 8
  Baseline AST: Abnormal | 0
  Post-Injection AST: number analyzed (Participants) | 5
  Post-Injection AST: Normal | 5
  Post-Injection AST: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Alkaline Phosphatase values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Alkaline Phosphatase values were normal
Statistical Analysis 2: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection ALT values. The values were categorized as Normal or Abnormal; p = 0.219, McNemar — The threshold for statistical significance was p = 0.05
Statistical Analysis 3: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection AST values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the AST values were normal

14. Secondary Outcome: Clinically Significant Change in White Blood Cell Count (WBC)
Description: White blood cell count measured in WBC/mm3 blood. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: All patients were scheduled to undergo complete blood count (CBC). Three patients did not undergo post-injection CBC due to various issues (IV or blood hemolysis).
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline WBC: Normal | 6
  Baseline WBC: Abnormal | 2
  Post-Injection WBC: number analyzed (Participants) | 5
  Post-Injection WBC: Normal | 4
  Post-Injection WBC: Abnormal | 1
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection WBC values. The values were categorized as Normal or Abnormal; p = 0.687, McNemar — The threshold for statistical significance was p = 0.05

15. Secondary Outcome: Clinically Significant Change in Hemoglobin (Hgb)
Description: Hgb measured in g/dL. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Hemoglobin: Normal | 7
  Baseline Hemoglobin: Abnormal | 1
  Post-Injection Hemoglobin: number analyzed (Participants) | 5
  Post-Injection Hemoglobin: Normal | 4
  Post-Injection Hemoglobin: Abnormal | 1
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Hemoglobin values. The values were categorized as Normal or Abnormal; p = 0.375, McNemar — The threshold for statistical significance was p = 0.05

16. Secondary Outcome: Clinically Significant Change in Hematocrit (Hct)
Description: Hct measured in %. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Hematocrit: Normal | 6
  Baseline Hematocrit: Abnormal | 2
  Post-Injection Hematocrit: number analyzed (Participants) | 5
  Post-Injection Hematocrit: Normal | 2
  Post-Injection Hematocrit: Abnormal | 3
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Hematocrit values. The values were categorized as Normal or Abnormal; p = 1.000, McNemar — The threshold for statistical significance was p = 0.05

17. Secondary Outcome: Clinically Significant Change in Platelets
Description: Platelets measured in platelets/mm3 blood. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline Platelets: Normal | 8
  Baseline Platelets: Abnormal | 0
  Post-Injection Platelets: number analyzed (Participants) | 5
  Post-Injection Platelets: Normal | 5
  Post-Injection Platelets: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection Platelets values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the Platelets values were normal

18. Secondary Outcome: Clinically Significant Change in Red Blood Cell Count (RBC)
Description: RBC measured in million/mm3. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline RBC: Normal | 7
  Baseline RBC: Abnormal | 1
  Post-Injection RBC: number analyzed (Participants) | 5
  Post-Injection RBC: Normal | 4
  Post-Injection RBC: Abnormal | 1
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection RBC values. The values were categorized as Normal or Abnormal; p = 0.375, McNemar — The threshold for statistical significance was p = 0.05

19. Secondary Outcome: Clinically Significant Change in Mean Corpuscular Volume (MCV)
Description: MCV measured in µm3. Values outside of laboratory range in comparison to baseline or >20% difference from baseline values.
Time Frame: 6 hours from 68Ga-Galmydar injection
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Dosimetry Group
Number analyzed (Participants) | 8
Participants
  Baseline MCV: Normal | 8
  Baseline MCV: Abnormal | 0
  Post-Injection MCV: number analyzed (Participants) | 5
  Post-Injection MCV: Normal | 5
  Post-Injection MCV: Abnormal | 0
Statistical Analysis 1: Comparison: Dosimetry Group; Test type: Equivalence — A McNemar test was performed between baseline and post-injection MCV values. The values were categorized as Normal or Abnormal; The McNemar test requires at least one participant for each outcome (Normal or Abnormal). Thus, no p-value was computed because all of the MCV values were normal

ADVERSE EVENTS:
Time Frame: 14 days after participant received injection of radiotracer
Description: Study staff contacted participants by phone following the administration of [68Ga]Galmydar to confirm the subject's well-being and to ascertain if an adverse event occurred post-imaging procedures. Subjects received a phone call within 2-3 days and at 5-7 days or as late as 14 days post [68Ga]Galmydar injection.
Arm/Group | Dosimetry Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/82/NCT05280782/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/82/NCT05280782/ICF_001.pdf